CLINICAL TRIAL: NCT01170468
Title: Does Vitamin D Reduce Risk of Developing Type II DM in Prediabetics? A Double Blind Randomized Controlled Trial
Brief Title: Does Vitamin D Reduce Risk of Developing Type II DM in High Risk Individuals
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: inadequate enrollement
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Muhammad Maher Hammami, Chairman, Department of Clinical Studies & Empirical Ethics, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RAC 2101040
Record Dates: First submitted 2010-07-25; First posted 2010-07-27 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Prediabetics; DM; vitamin D
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3 5000 IU daily
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 5000 IU orally, daily for 2 years
  Other Names: cholecalciferol
  Arms: Vitamin D3
Drug: Placebo — Placebo orally, daily for 2 years
  Arms: Placebo

SUMMARY:
Both vitamin D deficiency and type II DM/prediabetes are highly prevalent. Vitamin D status has been negatively associated with the presence of type II DM and glycemic control. A cause-effect relationship between vitamin D deficiency and the development of type II DM has not been established.

The investigators plan to conduct a 2 year, double blind, randomized, placebo controlled trial on the effect of vitamin D3 supplement on the incidence of type II DM in high risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults living in Riyadh area with impaired fasting glucose or/and impaired glucose tolerance (prediabetics) and total 25 OH vitamin D level between 10-30 nmol/l
* Who consume no more than one serving of milk/day
* Do not take vitamin supplement
* Habitually have less than 10 hour of sun exposure per week
* Don't suffer from granulomatus conditions, liver disease, kidney disease, or diabetes
* Don't take anticonvulsants, barbiturates, steroids, or antidiabetic medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01-15 (Actual); Study Completion 2014-01-15 (Actual)

PRIMARY OUTCOMES:
The incidence of DM | 2 years
  Development of DM diagnosed by glucose levels, fasting and/or 2-hour post 75 mg glucose challenge.

SECONDARY OUTCOMES:
slope of fasting glucose level | 2 years
slope of 2-hour post challenge glucose level | 2 years
area under the curve of BP | 2 years
area under the curve of weight | 2 years
area under the curve of 25 OH vitamin D level | 2 years
fasting insulin to glucose ratio | 2 years
incidence of hypercalcemia | 2 years
incidence of hypercalciuria | 2 years
time to develop DM | 2 years
  Development of DM diagnosed by glucose levels, fasting and/or 2-hour post 75 mg glucose challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Hammami, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia